CLINICAL TRIAL: NCT07355439
Title: The Effect of Positioning Duration on Pressure Injury Risk in Intensive Care Patients
Brief Title: Positioning Duration and Pressure Injury Risk
Acronym: PIP-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEMA ŞAHİNER (Other)
Collaborators: Bartin State Hospital (Other Government)
Responsible Party: Sponsor-Investigator, SEMA ŞAHİNER, graduate student, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-SBB-0140
Record Dates: First submitted 2025-12-16; First posted 2026-01-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pressure Injury; Risk Assessment
Keywords: pressure ınjury; moisture; position duration; intensive care unit; temperature
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: 82 patients will be divided into 2 groups. One group will have their position changed every hour, and the other group every two hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Position changes will be implemented at 1-hour intervals.
  Interventions: Behavioral: Position Change - 1 Hour
- control group (Active Comparator): Position changes will be implemented at 2-hour intervals.
  Interventions: Behavioral: Position Change - 2 Hours

INTERVENTIONS:
Behavioral: Position Change - 1 Hour — Patient positions will be changed at 1-hour intervals.
  Arms: experimental group
Behavioral: Position Change - 2 Hours — Patient positions will be changed at 2-hour intervals.
  Arms: control group

SUMMARY:
This research aims to investigate the effect of positioning times on the risk of pressure injury in critically ill patients.

DETAILED DESCRIPTION:
Pressure injuries, considered an indicator of quality of care, remain a significant concern today. They are a health problem that reduces the patient's quality of life, complicates the treatment process, and significantly increases costs. Immobility is one of the main risk factors for pressure injury development. In healthy individuals, discomfort occurs in an area subjected to pressure for a long enough period to cause ischemia, and the person changes their position via the afferent sensorimotor feedback system. Fewer than 20 movements per night significantly increase the risk of ulcer development. The factor causing ulcer formation is the inability of the individual to relieve the pressure applied to the tissue. Patients with limited mobility cannot change their body position on their own, and tissue perfusion is impaired in pressure-exposed areas, facilitating ulcer formation. Both the intensity and duration of pressure affect the effect. High pressure causes pressure to build up quickly, while the longer the pressure, the greater the risk of pressure buildup. In individuals at high risk of pressure injuries, frequent position changes are a primary policy for preventing pressure injuries. Experimental studies show that irreversible ischemia occurs when pressure is applied continuously for two hours or longer. The best method for reducing pressure in patients is repositioning. The literature indicates that while pressure injuries cannot be completely prevented, their incidence can be significantly reduced through evidence-based practices, particularly through assessment of at-risk patients, appropriate early nursing interventions, and preventive measures. Advances in the early detection of pressure injuries have been reported in the literature and primarily involve measuring inflammatory markers in anatomical regions to capture the first signs of tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* - If the patient is conscious, they must volunteer to participate in the study.
* For unconscious patients, a first-degree relative (mother, father, spouse, child) must agree to participate in the study.
* The patient's dependency level score on the Barthel Activities of Daily Living Index must be 90 or below (moderately dependent, severely dependent, completely dependent).
* The patient must not have developed a pressure injury.
* The patient must be meeting their daily calorie needs as determined by the nutrition team.
* There must be no contraindications to turning the patient to any side.
* Patients who are at low risk according to the pressure injury scale (15 points or above according to the Braden Risk Assessment Scale).
* The patient must not have an acute neurological problem.
* Patients with a GCS score above 7.

Exclusion Criteria:

* - If the patient is conscious, they do not consent to participate in the study.
* For unconscious patients, their first-degree relative does not consent to participate in the study.
* Patients with a Barthel Activities of Daily Living Index score above 90 (mildly dependent, fully independent).
* The patient has an existing pressure injury.
* The patient is not meeting their daily calorie needs as determined by the nutrition team.
* There is a contraindication to turning the patient to any side.
* Patients with moderate to high risk according to the pressure injury scale (score below 15 according to the Braden Risk Assessment Scale).
* The patient has an acute neurological problem.
* Patients with a GCS score of 7 or below.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Skin Integrity Changes | Recording body temperature by measuring it with a body temperature measurement device every 24 hours for 72 hours.
  Evaluation of changes in body temperature as a risk factor for pressure injury.
Skin Integrity Changes | Body moisture will be assessed and documented every 24 hours over a 72-hour period using a body moisture measurement device.
  Evaluation of changes in body moisture level as a risk factor for pressure injury
Skin Integrity Changes | Whether changes in skin appearance, such as bruising, occur will be assessed and recorded through observation every 24 hours over a 72-hour period.
  Assessment of the occurrence of changes in skin appearance, such as bruising, considered as risk factors for pressure injury.
Skin Integrity Changes | The presence of changes in skin appearance, such as edema, will be assessed and recorded through observation at 24-hour intervals over a 72-hour period.
  Assessment of the occurrence of changes in skin appearance, such as edema, considered as risk factors for pressure injury.
Skin Integrity Changes | The presence of changes in skin appearance, such as redness, will be assessed and recorded through observation at 24-hour intervals over a 72-hour period.
  Assessment of the occurrence of changes in skin appearance, such as redness, considered as risk factors for pressure injury.

SECONDARY OUTCOMES:
Braden Risk Assessment Score | Evaluations will be conducted and documented at 24-hour intervals over a 72-hour period using the scale.
  Pressure injury risk will be quantitatively assessed using the Braden Pressure Ulcer Risk Assessment Scale, which consists of six subdimensions: sensory perception, moisture, activity, mobility, nutrition, and friction/shear. Total scores range from 6 to 23, with decreasing scores over the assessment period indicating an increased risk of pressure ulcer development.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartin University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In this study, individual patient data was used in an anonymized form and will not be shared with third parties in accordance with the principles of patient privacy and the protection of personal data.

REFERENCES:
- [Background] Esra ÖZKAN, Kemal TURHAN, The Effect of Position Time on the Formation of Pressure Ulcer in Bedridden Patients, Turkiye Klinikleri J Nurs Sci. 2019;11(3):246-54.
- See also: NATIONAL PRESSURE ULCER ADVISORY PANEL — https://npiap.com/